CLINICAL TRIAL: NCT01866540
Title: The Systemic And Local Immune Response To Intranasal Influenza Vaccination
Brief Title: Immune Response To Intranasal Influenza Vaccination
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Rebecca Cox, Professor, University of Bergen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LAIV-tonsilsv2 Version 2; 2012-002848-24 (EudraCT Number)
Record Dates: First submitted 2012-10-22; First posted 2013-05-31 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Tonsillitis, Hypertrophy
Keywords: influenza, LAIV, immune response
MeSH Terms: conditions — Tonsillitis; Hypertrophy; Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluenz vaccine (Experimental): LAIV vaccine
  Interventions: Drug: FLUENZ

INTERVENTIONS:
Drug: FLUENZ — live attenuated influenza vaccine
  Other Names: FLUMIST

SUMMARY:
This research during the last decade has focused on the kinetics of the systemic and local immune response to parenteral influenza vaccine in humans. The investigators have shown that normally high numbers of influenza specific antibody secreting cells (ASC) are present in the nasal mucosa of healthy adults but upon parenteral vaccination the numbers remain stable. However, a rapid transient increase in specific ASC is observed in the tonsils and peripheral blood after parenteral vaccination. In the tonsils, this is associated with a significant decrease in both naïve/effector (CD45RA+) and memory (CD45RO+) CD4+ cells upon vaccination. In this study the investigators will extend our work to investigate the characteristics of influenza-specific T- and B-cells induced locally and systemically after intranasal vaccination in man.

DETAILED DESCRIPTION:
The clinical trial will be an open study. All subjects eligible for tonsillectomy at Haukeland University Hospital within the specified age range (children: 2 to less than 18 years old and adults >18-59 years old) will receive an invitation to join the study. The primary endpoints of the trial are the evaluation of the systemic and local immune response after live attenuated influenza vaccine. The vaccine specific immune response will be assessed through the induction of specific local and systemic antibody and cellular immune responses, and analyses of the epitopes to which the response is directed. Furthermore the capacity of the vaccine to elicit cross reactive and long lasting immunity will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (age range ≥2 and <18 years old) or adults (>18-59 years old) as concluded from the medical history, physical examination, and clinical judgment) scheduled for tonsillectomy ;
* Signed informed consent from the subject or both parents/ both guardians and from subjects aged 12 years and older;
* Subjects or guardians able to understand and comply with the study protocol and complete the Adverse Event Form:
* Subjects able to attend the scheduled visits.

Exclusion Criteria:

* Persons with a history of anaphylaxis or serious reactions to any vaccine;
* Person with known hypersensitivity to any of the vaccine components (e.g. gelatin, gentamicin, eggs or egg proteins (e.g. ovalbumin);
* Persons who are pregnant
* Persons who have had a temperature >38oC during the previous 72 hours;
* Persons who have had an acute respiratory infection during the last 7 days;
* Persons who are clinically immunodeficient due to conditions or immunosuppressive therapy such as: acute and chronic leukaemias; lymphoma; symptomatic HIV infection; cellular immune deficiencies; and high-dose corticosteroids;
* Persons with severely immunocompromised family members;
* Persons with severe asthma or active wheezing.

Ages: 2 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-10-01; Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
evaluation of the systemic and local immune response after live attenuated influenza vaccine. | 1 year
  Measurement of systemic and local immune responses in immunological assays

OTHER OUTCOMES:
Influenza specific responses | 31.12.2015
  induction of specific local and systemic antibody and cellular immune responses, and analyses of the epitopes to which the response is directed. Furthermore the capacity of the vaccine to elicit cross reactive and long lasting immunity will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Hans Jørgen Aarstad, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Result] Lartey S, Zhou F, Brokstad KA, Mohn KG, Slettevoll SA, Pathirana RD, Cox RJ. Live-Attenuated Influenza Vaccine Induces Tonsillar Follicular T Helper Cell Responses That Correlate With Antibody Induction. J Infect Dis. 2020 Jan 1;221(1):21-32. doi: 10.1093/infdis/jiz321. PMID 31250024
- [Result] Islam S, Zhou F, Lartey S, Mohn KGI, Krammer F, Cox RJ, Brokstad KA. Functional immune response to influenza H1N1 in children and adults after live attenuated influenza virus vaccination. Scand J Immunol. 2019 Oct;90(4):e12801. doi: 10.1111/sji.12801. Epub 2019 Sep 2. PMID 31269273
- [Result] Islam S, Mohn KG, Krammer F, Sanne M, Bredholt G, Jul-Larsen A, Tete SM, Zhou F, Brokstad KA, Cox RJ. Influenza A haemagglutinin specific IgG responses in children and adults after seasonal trivalent live attenuated influenza vaccination. Vaccine. 2017 Oct 9;35(42):5666-5673. doi: 10.1016/j.vaccine.2017.08.044. Epub 2017 Sep 9. PMID 28899626
- [Result] Mohn KGI, Zhou F, Brokstad KA, Sridhar S, Cox RJ. Boosting of Cross-Reactive and Protection-Associated T Cells in Children After Live Attenuated Influenza Vaccination. J Infect Dis. 2017 May 15;215(10):1527-1535. doi: 10.1093/infdis/jix165. PMID 28368530
- [Result] Manenti A, Tete SM, Mohn KG, Jul-Larsen A, Gianchecchi E, Montomoli E, Brokstad KA, Cox RJ. Comparative analysis of influenza A(H3N2) virus hemagglutinin specific IgG subclass and IgA responses in children and adults after influenza vaccination. Vaccine. 2017 Jan 3;35(1):191-198. doi: 10.1016/j.vaccine.2016.10.024. Epub 2016 Oct 24. PMID 27789145
- [Result] Mohn KG, Brokstad KA, Pathirana RD, Bredholt G, Jul-Larsen A, Trieu MC, Lartey SL, Montomoli E, Tondel C, Aarstad HJ, Cox RJ. Live Attenuated Influenza Vaccine in Children Induces B-Cell Responses in Tonsils. J Infect Dis. 2016 Sep 1;214(5):722-31. doi: 10.1093/infdis/jiw230. Epub 2016 May 30. PMID 27247344
- [Result] Panapasa JA, Cox RJ, Mohn KG, Aqrawi LA, Brokstad KA. The expression of B & T cell activation markers in children's tonsils following live attenuated influenza vaccine. Hum Vaccin Immunother. 2015;11(7):1663-72. doi: 10.1080/21645515.2015.1032486. PMID 26148331
- [Result] Mohn KG, Bredholt G, Brokstad KA, Pathirana RD, Aarstad HJ, Tondel C, Cox RJ. Longevity of B-cell and T-cell responses after live attenuated influenza vaccination in children. J Infect Dis. 2015 May 15;211(10):1541-9. doi: 10.1093/infdis/jiu654. Epub 2014 Nov 25. PMID 25425696
- [Result] Pidelaserra Marti G, Isdahl Mohn KG, Cox RJ, Brokstad KA. The influence of tonsillectomy on total serum antibody levels. Scand J Immunol. 2014 Nov;80(5):377-9. doi: 10.1111/sji.12213. No abstract available. PMID 25039393
- See also: Influenza Centre — http://www.influensasenteret.no